CLINICAL TRIAL: NCT04551079
Title: A Randomized, Double-Blind, Placebo-Controlled, 3-Period Crossover Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of Oral TAK-994 in an Acute Sleep Phase Delay Paradigm in Healthy Male Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics (PK) of Oral TAK-994 in an Acute Sleep Phase Delay Paradigm in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: TAK-994-1503; U1111-1256-7132 (Registry Identifier: WHO)
Record Dates: First submitted 2020-09-11; First posted 2020-09-16 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAK-994 Dose A+ Placebo + TAK-994 Dose B (Experimental): TAK-994 Dose A tablets, orally, on Days 1 and 2 of Treatment Period 1, followed by TAK-994 placebo-matching tablets, orally, on Days 1 and 2 of Treatment Period 2, further followed by TAK-994 Dose B tablets, orally, on Days 1 and 2 of Treatment Period 3. A Washout Period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: TAK-994; Drug: Placebo
- TAK-994 Dose B + TAK-994 Dose A + Placebo (Experimental): TAK-994 Dose B tablets, orally, on Days 1 and 2 of Treatment Period 1, followed by TAK-994 Dose A tablets, orally, on Days 1 and 2 of Treatment Period 2, further followed by TAK-994 placebo-matching tablets, orally, on Days 1 and 2 of Treatment Period 3. A Washout Period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: TAK-994; Drug: Placebo
- Placebo + TAK-994 Dose B+ TAK-994 Dose A (Experimental): TAK-994 placebo-matching tablets, orally, on Days 1 and 2 of Treatment Period 1, followed by TAK-994 Dose B tablets orally, on Days 1 and 2 of Treatment Period 2, further followed by TAK-994 Dose A tablets, orally, on Days 1 and 2 of Treatment Period 3. A Washout Period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: TAK-994

INTERVENTIONS:
Drug: TAK-994 — TAK-994 tablets.
Drug: Placebo — TAK-994 placebo-matching tablets.
  Arms: TAK-994 Dose A+ Placebo + TAK-994 Dose B; TAK-994 Dose B + TAK-994 Dose A + Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of TAK-994 and to determine the effect of TAK-994 (compared to placebo) on sleepiness, as measured by mean sleep latency on the maintenance of wakefulness Test (MWT), in an acute sleep phase delay paradigm in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-994. The study will evaluate the safety/tolerability, PD, and PK of TAK-994 in an acute sleep phase delay paradigm in healthy participants.

The study will enroll up to approximately 18 healthy participants. Participants will be randomly assigned to 1 of the 3 treatment sequences which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* TAK-994 Dose A + Placebo + TAK-994 Dose B
* TAK-994 Dose B + TAK-994 Dose A + Placebo
* Placebo + TAK-994 Dose B + TAK-994 Dose A

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 10 weeks. Participants will be followed up remotely on Day 7 after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Be a current nonsmoker who has not used tobacco- or nicotine-containing products (example, nicotine patch) for at least 6 months prior to the first dose of study drug.
2. Have regular sleep-wake habits (example, routinely spending 6.5 to 8 hour sleeping nightly, not oversleeping by more than 3 hour on weekends [that is, total sleep not more than 11 hour]) as determined by investigator interviews and confirmed in 5-day actigraphy records and regularly fall asleep between 9:30 PM and 12:00 AM.

Exclusion Criteria:

1. Have a positive alcohol or drug screen or a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce] per day).
2. Have excessive sleepiness, defined by a self-reported Epworth Sleepiness Scale (ESS) score at screening greater than (>) 10; irregular work hours; or routine night-shift work within 1 month before randomization.
3. Have a prior history of or currently is experiencing any known/suspected sleep disorder (including obstructive sleep apnea and restless leg syndrome), any disorder associated with excessive daytime sleepiness (EDS), or any diagnosis interfering with assessment of sleepiness.
4. At the time of screening, be receiving treatment with nasal/oronasal positive airway pressure for any reason.
5. Have abnormal findings on the initial polysomnography conducted on Day -1 (check-in) of the first treatment period.
6. Have traveled across 2 or more time zones within the 2 weeks before screening.
7. Have caffeine consumption of more than 400 milligram (mg)/day for 2 weeks before screening (1 serving of coffee is approximately equivalent to 120 mg of caffeine).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Experience at Least 1 Treatment Emergent Adverse Event (TEAE) During the Study | From first dose of the study drug up to Day 7 after the last dose of study drug on Day 2 in Treatment Period 3 (up to Day 27)
Number of Participants who Meet the Markedly Abnormal Value for Safety Laboratory Tests at Least Once Postdose During the Study | From first dose of the study drug up to Day 7 after the last dose of study drug on Day 2 in Treatment Period 3 (up to Day 27)
Number of Participants who Meet the Markedly Abnormal Value for Vital Sign Measurements at Least Once Postdose During the Study | From first dose of the study drug up to Day 7 after the last dose of study drug on Day 2 in Treatment Period 3 (up to Day 27)
Number of Participants who Meet the Markedly Abnormal Value for Safety Electrocardiogram (ECG) Parameters at Least Once Postdose During the Study | From first dose of the study drug up to Day 7 after the last dose of study drug on Day 2 in Treatment Period 3 (up to Day 27)
Mean Sleep Latency Over Four Maintenance of Wakefulness Test (MWT) Sessions After Initial Dosing | Up to 8 hours after initial dosing in each treatment period
  MWT is a validated objective measure that evaluates a person's ability to remain awake under soporific conditions for a defined period of time. Tendency to fall asleep is measured via electroencephalography-derived sleep latency. Mean sleep latency: mean time to sleep onset, over 4 MWT sessions (at approximately 2, 4, 6, and 8 hours after initial dosing).

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for TAK-994 | Days 1 and 2: Pre-dose and at multiple time points (up to 10 hours) post-dose
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-994 | Days 1 and 2: Pre-dose and at multiple time points (up to 10 hours) post-dose
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-994 | Days 1 and 2: Pre-dose and at multiple time points (up to 10 hours) post-dose
Change From Baseline in Mean Karolinska Sleepiness Scale (KSS) Score | Baseline up to 8.75 hours after initial dosing in each treatment period
  The KSS is a 10-item, Likert-type rating scale for assessing subjective sleepiness. This participant self-rating scale measures the subjective level of sleepiness at the time of administration.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Clinilabs Drug Development Corporation, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.